CLINICAL TRIAL: NCT04459429
Title: Effect of Cannula Size on Peripheral Oxygen Saturation During Nasal High Flow Therapy in Neonates With Respiratory Distress
Brief Title: Effect of Cannula Size on Oxygen Saturation During Nasal High Flow Therapy in Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erebouni Medical Center (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Principal Investigator, Pavel Mazmanyan, Professor, Erebouni Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Erebouni01Neonatal
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: RDS - Infants; TTN
Keywords: RDS; TTN; Nasal High Flow Therapy; Newborn
MeSH Terms: conditions — RDS - infants

STUDY DESIGN:
Intervention Model Description: Randomized crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NHF by smaller cannula (Experimental): Nasal High Flow will be applied at 8 L/min (AIRVO 2) through the smaller cannula
  Interventions: Device: Change of cannula size
- NHF by larger cannula (Experimental): Nasal High Flow will be applied at 8 L/min (AIRVO 2) through the larger cannula
  Interventions: Device: Change of cannula size

INTERVENTIONS:
Device: Change of cannula size — During nasal High Flow Therapy with fixed flow of 8 l/min, the cannula size will be changed from smaller-to-larger or larger-to-smaller

SUMMARY:
Treatment with nasal high flow therapy (NHF) is an increasingly popular method of respiratory support in newborns.

Safe and effective use of NHF requires selection of an appropriate nasal prong-to-nares ratio because leak can influence the delivered pressure.

To the best of our knowledge, this is the first study to investigate the effect of using different NHF cannula size on peripheral oxygen saturation in newborns with respiratory distress.

DETAILED DESCRIPTION:
NHF will be applied at 8 L/min using the AIRVO 2 through smaller and larger Optiflow nasal cannula. The study will have a randomized crossover design. The larger or smaller cannula size will be applied as the first intervention during each experiment. During each experiment, if the larger cannula is applied first, then the smaller cannula will be applied second and if the smaller cannula is applied first, then the larger cannula will be applied second. Each experiment will last for 1.5 hour.

* During baseline, supplemental oxygen will be added during NHF therapy to keep SpO2 in normal ranges (90%-94%). When the SpO2 has stabilized then the level of supplemental oxygen will be set for the entire experiment unless there is a significant change in SpO2 as determined by the attending consultant.
* There will be three consecutive 30-min periods of recording during each experiment and each experiment will last approximately 1.5 hour.
* Ventilation will be assessed by Respiratory Inductance Plethysmography (Respitrace) and transcutaneous carbon dioxide and oxygen.
* Recordings will be made using ADInstruments Powerlab and Labchart software with video recording of the patient.
* Routine measurement of heart rate, respiratory rate and oxygen saturations will be performed as per standard neonatal practice.

The researcher is an experienced neonatal consultant who will be directly observing the baby throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Term and near term newborns with respiratory distress receiving treatment with NHF
2. ≤ 48 hours old
3. FiO2 ≥ 0,4
4. Written parental informed consent

Exclusion Criteria:

1. Infants who are clinically unstable and unsuitable for non-invasive respiratory support as judged by consultant clinician (meet nHF failure criteria).
2. Known major upper airway, lower respiratory tract, cardiac or gastrointestinal tract anomaly
3. A parent has not given written informed consent to their baby's participation.
4. Prior intubation and/or surfactant administration
5. Known or suspected hypoxic ischemic encephalopathy

Ages: 1 Hour to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2020-12-24 (Actual)

PRIMARY OUTCOMES:
Peripheral oxygen saturation (SpO2 ) | 1.5 hour
  The difference in SpO2 between the period of using the larger cannula versus the smaller cannula

SECONDARY OUTCOMES:
inspiratory effort | 1.5 hour
  The difference in inspiratory effort between the period of using the larger cannula versus the smaller cannula
Respiratory rate | 1.5 hour
  The change in respiratory rate between the period of using the larger cannula versus the smaller cannula
Relative minute ventilation | 1.5 hour
  The difference in relative minute ventilation (inspiratory effort x respiratory rate) during the periods of using the larger cannula versus smaller cannula
Pulse rate | 1.5 hour
  The difference in pulse rate between the period of using the larger cannula versus the smaller cannula
Transcutaneous carbon dioxide | 1.5 hour
  The difference in TcCO2 between the period of using the larger cannula versus the smaller cannula
Transcutaneous oxygen | 1.5 hour
  The difference in TcO2 between the period of using the larger cannula versus the smaller cannula

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Mazmanyan, MD, PhD, Principal Investigator — Erebouni Medical Center
Locations (1):
- Erebouni Medical Center Maternity, Yerevan, Armenia

IPD SHARING:
Plan to Share IPD: No
There is currently no intent to share individual data with other researchers.